CLINICAL TRIAL: NCT05838170
Title: A Phase 2, Randomized, Double-Blind, Vehicle-Controlled, Parallel-Group Study Evaluating the Safety, Tolerability, and Efficacy of TP-04 in Participants With Papulopustular Rosacea
Brief Title: Study of TP-04 in Participants With Papulopustular Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tarsus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRS-016
Record Dates: First submitted 2023-03-13; First posted 2023-05-01 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Papulopustular Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Intervention Model Description: The investigational product (Lotilaner Gel, 2.0% [TP-04]) or vehicle control gel will be applied topically on the face twice daily (BID) during the study.
  Participants will be randomized to a 2:1 ratio at baseline to apply Lotilaner Gel, 2.0% (TP-04) or vehicle control gel on the face BID for 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind, Vehicle-Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lotilaner Gel, 2.0% (TP-04) (Experimental): Participants will be randomized to a 2:1 ratio at baseline to apply Lotilaner Gel, 2.0% (TP-04) on the face BID for 12 weeks.
  Interventions: Drug: Lotilaner Gel, 2.0%
- Vehicle-Controlled (Placebo Comparator): Participants will be randomized to a 2:1 ratio at baseline to apply vehicle control gel on the face BID for 12 weeks.
  Interventions: Other: Vehicle control gel

INTERVENTIONS:
Drug: Lotilaner Gel, 2.0% — Lotilaner Gel, 2.0% (TP-04) is an aqueous gel formulation of lotilaner, a member of the isoxazoline family of compounds and parasiticide that selectively inhibits parasite-specific gamma-aminobutyric acid (GABA)-gated chloride channels (GABA-Cls).
  Other Names: TP-04
  Arms: Lotilaner Gel, 2.0% (TP-04)
Other: Vehicle control gel — Aqueous gel
  Other Names: Vehicle Gel
  Arms: Vehicle-Controlled

SUMMARY:
This study is being done to evaluate the safety, tolerability, and efficacy of the study drug, TP-04, in participants with papulopustular rosacea (PPR).

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-blind, parallel-group, vehicle-controlled study evaluating the safety, tolerability, and efficacy of Lotilaner Gel, 2.0% (TP-04) applied BID for 12 weeks in participants with moderate to severe PPR.

ELIGIBILITY:
Inclusion criteria:

1. Participant is willing to participate and is capable of giving informed consent. Note: Consent must be obtained prior to any study-related procedures.
2. Male or female participant aged 18 to 59 years, inclusive, at the time of consent.
3. Participant has at least a 6-month history of PPR at the screening visit (information obtained from medical chart or participant's physician, or directly from the participant).
4. Participant has moderate or severe PPR, as defined by an IGA score of 3 (moderate) or 4 (severe) at the screening and Day 1 visits.
5. Participant has 20 to 70 inflammatory lesions (papules and/or pustules) and no more than 2 nodules (defined as a lesion ˃ 5 mm in diameter) on the face at the screening and Day 1 visits.
6. Participant has moderate or severe persistent erythema associated with PPR, as defined by a CEA score of 3 (moderate) or 4 (severe) at the screening and Day 1 visits.
7. Participant has SSSB1 > 5 D/cm² or SSSB2 > 10 D/cm² at the screening and Day 1 visits.
8. Female participant of childbearing potential has had a negative serum pregnancy test at screening and a negative urine pregnancy test at Day 1.
9. For female participant of childbearing potential involved in any sexual intercourse that could lead to pregnancy: the participant must agree to use a highly effective contraceptive method from at least 4 weeks prior to Day 1 until at least 6 months after the last study product application. Highly effective contraceptive methods include hormonal contraceptives (eg, combined oral contraceptive, patch, vaginal ring, injectable, or implant), intrauterine devices or intrauterine systems, vasectomized partner(s) (provided his vasectomy was performed ≥ 4 months prior to screening), tubal ligation or double barrier methods of contraception (eg, male condom with cervical cap, male condom with diaphragm, and male condom with contraceptive sponge) in conjunction with spermicide.
10. For male participant involved in any sexual intercourse that could lead to pregnancy, participant must agree to use one of the highly effective contraceptive methods listed in Inclusion Criterion #9, from Day 1 until at least 6 months after the last study product application. If the female partner of a male participant use any of the hormonal contraceptive methods listed above, this contraceptive method should be used by the female partner from at least 4 weeks before Day 1 until at least 6 months after the last study product application.
11. For participant who uses makeup, facial moisturizers, creams, lotions, cleansers, and/or sunscreens, participant has used the same product brands/types for a minimum period of 2 weeks prior to Day 1, agrees not to change brand/type or frequency of use throughout the study, and agrees not to use makeup, facial moisturizers, creams, lotions, cleansers, and/or sunscreens prior to study visits. Participants will be instructed not to apply these products on the treated areas within approximately 30 minutes before and after study product application.
12. Participant is willing to limit or avoid known personal triggers of rosacea (eg, spicy foods, consumption of alcoholic beverages, extended intentional sun exposure, tanning beds, sauna, etc) for the duration of the study.
13. Participants must be willing to comply with all study procedures and must be available for the duration of the study.

Exclusion criteria:

1. Participant is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
2. Participant has rosacea conglobata, rosacea fulminans, perioral dermatitis, facial erythrosis other than rosacea, corticosteroid-induced rosacea, facial keratosis pilaris, facial seborrheic dermatitis, acute lupus erythematosus, chronic recurring facial acne vulgaris, isolated rhinophyma, or plaque- like facial edema or with ocular rosacea (blepharitis, keratitis) requiring or likely to require systemic treatment.
3. Participant has a history of skin disease, presence of a skin condition, scarring, excessive facial hair, tattoos, or other facial characteristics (eg, actinic damage) that could, in the opinion of the investigator, interfere with study assessments.
4. Participant has any clinically significant medical condition or physical/laboratory/ECG/vital signs abnormality that would, in the opinion of the investigator, put the participant at undue risk or interfere with interpretation of study results.
5. Participant has a history of cancer or lymphoproliferative disease within 5 years prior to Day 1. Participants with successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix are not to be excluded.
6. Participant has a known history of chronic infectious disease (eg, hepatitis B, hepatitis C, or human immunodeficiency virus [HIV]).
7. Participant has used oral retinoids (eg, isotretinoin) within 52 weeks prior to Day 1 or high-dose vitamin A (> 10,000 IU/day) within 26 weeks prior to Day 1.
8. Participant has received any marketed or investigational biological agent within 12 weeks or 5 half-lives (whichever is longer) prior to Day 1.
9. Participant has received hormonal therapy that is not on a stable dose and frequency for at least 12 weeks before Day 1 or that is not maintained throughout the study.
10. Participant has received photodynamic therapy, phototherapy with blue or red light, or laser therapy to the face within 8 weeks prior to Day 1.
11. Participant had a major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study.
12. Participant has used systemic immunosuppressants (eg, steroids, steroid injections, cyclosporine, methotrexate, mycophenolate mofetate) within 8 weeks prior to Day 1.
13. Participant had a facial procedure (eg, chemical peel, microdermabrasion) within 8 weeks prior to Day 1.
14. Participant has used systemic products that could affect PPR within 4 weeks prior to Day 1 (eg, oral antibiotics, ivermectin).
15. Participant is currently receiving a nonbiological investigational product or device or has received one within 4 weeks prior to Day 1.
16. Participant has used any narrow therapeutic index (NTI) drug metabolized by cytochrome P450 (CYP)2C8, CYP2C19, CYP2C9, or CYP2D6 within 4 weeks prior to Day 1 or may require using any NTI drug metabolized by CYP2C8, CYP2C19, CYP2C9, or CYP2D6 within 8 weeks after the last study product application.
17. Participant is exposed to excessive sunlight (eg, working outside), is planning a trip to a sunny climate, or has used tanning booths within 4 weeks prior to Day 1 or is not willing to minimize exposure to natural and artificial sunlight or weather extremes (wind or cold) during the study.
18. Participant has used topical products that could affect PPR within 2 weeks prior to Day 1 (eg, metronidazole, azealeic acid, topical minocycline, sulfacetamide, resorcinol, clindamycin, topical ivermectin, tea tree oil, dapsone, cannabidiol [CBD]-containing products, topical calcineurin inhibitors, benzyl peroxide, topical retinoid/retinol, alpha or beta hydroxy-acids, phosphodiesterase 4 [PDE4] inhibitors, topical Janus kinase [JAK] inhibitors, oxymetazoline, bromonidine).
19. Participant has used on the face an over-the-counter (OTC) or prescription topical medication for rosacea, including benzoyl peroxide, topical anti-inflammatory medications, corticosteroids, salicylic acid, α-hydroxy/glycolic, or antibacterial/antiseptic soap or wash within 2 weeks prior to Day 1.
20. Participant has a known or suspected allergy to Lotilaner Gel, 2.0% (TP-04) or any component of the investigational product.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
The incidence of treatment emergent adverse events from baseline | Week 1 through Week 12
  Incidence of local and systemic TEAEs while using Lotilaner Gel, 2.0% (TP-04) versus vehicle control gel from baseline
Changes from baseline in vital signs change in height in cm | Week 1 through Week 12
  Changes from baseline in vital signs change in height in cm while using Lotilaner Gel, 2.0% (TP-04) versus vehicle control gel
Changes from baseline in vital signs change in weight in kg | Week 1 through Week 12
  Changes from baseline in vital signs change in weight in kg while using Lotilaner Gel, 2.0% (TP-04) versus vehicle control gel
Changes from baseline in vtial signs change in systolic/diastolic blood pressure in mmHg | Week 1 through Week 12
  Changes from baseline in vital signs change in systolic/diastolic blood pressure in mmHg while using Lotilaner Gel, 2.0% (TP-04) versus vehicle control gel
Changes from baseline in vital signs change in pulse in beats per minute | Week 1 through Week 12
  Changes from baseline in vital signs change in pulse in beats per minute while using Lotilaner Gel, 2.0% (TP-04) versus vehicle control gel
Changes from baseline in vital signs change in respiratory rate in breaths per minute | Week 1 through Week 12
  Changes from baseline in vital signs change in respiratory rate in breaths per minute while using Lotilaner Gel, 2.0% (TP-04) versus vehicle control gel
Changes from baseline in vital signs change in temperature in Celsius | Week 1 through Week 12
  Changes from baseline in vital signs change in temperature in Celsius while using Lotilaner Gel, 2.0% (TP-04) versus vehicle control gel
Change from baseline in ECGs change in QRS interval in msec | Week 1 through Week 12
  Changes from baseline in ECGs change in QRS interval in msec while using Lotilaner Gel, 2.0% (TP-04) versus vehicle control gel
Changes from baseline in ECGs change in mean ventricular rate (beats/min) | Week 1 through Week 12
  Changes from baseline in ECGs change in mean ventricular rate (beats/min) while using Lotilaner Gel, 2.0% (TP-04) versus vehicle control gel
Changes in baseline in ECGs change in QTC interval in msec | Week 1 through Week 12
  Changes from baseline in ECGs change in QTC interval in msec while using Lotilaner Gel, 2.0% (TP-04) versus vehicle control gel
Changes in clinical chemistry laboratory assessments from baseline | Week 1 through Week 12
  Changes from baseline clinical chemistry laboratory values while using Lotilaner Gel, 2.0% (TP-04) versus vehicle control gel
Changes in hematology laboratory assessments from baseline | Week 1 through Week 12
  Changes from baseline hematology laboratory values while using Lotilaner Gel, 2.0% (TP-04) versus vehicle control gel
Local tolerability assessment ((0=none, 3=severe): dryness, scaling, erythema, burning/stinging; itching) | Week 1 through Week 12
  Evaluate local tolerability assessment ((0=none, 3=severe): dryness, scaling, erythema, burning/stinging; itching) of Lotilaner Gel, 2.0% (TP-04) versus vehicle control gel

SECONDARY OUTCOMES:
Improvement in Investigator Global Assessment (IGA) score (0=clear; 4=severe) | Week 1 through Week 12
  Proportion (%) of participants achieving ≥ 2-point improvement in IGA score to clear (0) or almost clear (1)
Facial Inflammatory lesion counts - absolute change from baseline | Week 1 through Week 12
  Absolute change from baseline in facial inflammatory lesion counts
Facial inflammatory lesion counts - percent change from baseline | Week 1 through Week 12
  Percent change from baseline in facial inflammatory lesion counts
Investigator Global Assessmen (IGA) Score (0=clear; 4=severe) - absolute change from baseline | Week 1 through Week 12
  Absolute change from baseline in IGA score
Clinician Erythema Assessment (CEA) Score (0=clear; 4=severe) - absolute change from baseline | Week 1 through Week 12
  Absolute change from baseline in CEA score
Pruritus Numeric Rating Scale (NRS) Score (0=no itch; 10= worst imaginable itch) - absolute change from baseline | Week 1 through Week 12
  Absolute change from baseline in worst pruritus NRS score
Worst Pain Numeric Rating Scale (NRS) Score (0=no pain; 10= worst imaginable pain) - absolute change from baseline | Week 1 through Week 12
  Absolute change from baseline in worst pain NRS score
Improvement in Worst Pruritus Numeric Rating Scale (NRS) Score (0=no itch; 10= worst imaginable itch) | Week 1 through Week 12
  Proportion (%) of participants achieving at least a 4-point reduction in worst pruritus NRS score (0= no itch; 10= worst imaginable itch)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Trevejo, MD, PhD, Study Director — Tarsus Pharmaceuticals, Inc.
Locations (5):
- Canada (5):
  - The Centre for Clinical Trials, Oakville, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Saint-Louis, Québec

IPD SHARING:
Plan to Share IPD: No